CLINICAL TRIAL: NCT02530203
Title: Spinal Cord Stimulation to Treat Post-operative Atrial Fibrillation
Acronym: SCS-PAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a change in medication guidelines it became practically impossible to recruit patients
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCS-PAF
Record Dates: First submitted 2015-05-11; First posted 2015-08-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Fibrillation
Keywords: post-operative atrial fibrillation; spinal cord stimulation; CABG
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional treatment (Other): Non interventional group, patients that belong to this arm will receive the conventional treatment for CABG and they will wear the Holter for 5 days.
  Interventions: Device: Holter Recording_ NEMon DR220 Holter Recorders
- Spinal Cord Stimulation System (Experimental): This group will receive the Spinal Cord Stimulation System and they will wear the Holter for 5 days.
  Interventions: Device: Spinal Cord Stimulation System; Device: Holter Recording_ NEMon DR220 Holter Recorders

INTERVENTIONS:
Device: Spinal Cord Stimulation System — High frequency stimulation using a catheter placed in the lumen of the spine to inhibit sympathetic outflow to the heart
  Other Names: (Medtronic External Neurostimulator Model 37022; Medtronic 1x8 Standard LZ Lead Model 3877; Medtronic MultiLead Trialing Cable MLTC Model 355531)
  Arms: Spinal Cord Stimulation System
Device: Holter Recording_ NEMon DR220 Holter Recorders — To measure primary endpoint and most of the secondary endpoints in all the patients enrolled in the study. The recording will start to before CABG procedure and will be stop at day 5.

SUMMARY:
Patients will be randomized to control and spinal cord stimulation arm (SCS) to investigate the effect of SCS on the occurrence of post-operative atrial fibrillation in the five days after surgery.

DETAILED DESCRIPTION:
Pre market single center clinical research feasibility study. Non blinded randomized controlled study. 52 patients undergoing CABG procedure will be enrolled and randomized into two different group (26 person each): the Spinal Cord Stimulation (SCS) and the control group. The first group will be implanted before the CABG procedure with a temporary SCS lead (5 days) while the second one will not. The lead will be connected to an external stimulator.

The day of the CABG surgery, before the scheduled procedure, the patients in the treatment group will be implanted with the SCS lead. CABG procedure follows the SCS lead implantation. SCS will be switched off before surgery.

After the CABG procedure, all patients will be hospitalized for minimally five days at the end of which they will be discharged. The Primary Endpoint data will be collected from the day of CABG procedure (Day-0) until Day-5. SCS lead will be removed on Day-5.

1-week follow up visit will be performed one week after discharge. End-points will be evaluated at various time before, during and after surgery. In both groups arrhythmic episodes for primary and secondary endpoints will be recorded via a Holter monitor (recording 5 days continuously).

ELIGIBILITY:
Inclusion Criteria:

1. Patients which will be subjected to an OFF-pump CABG procedure
2. More than 18 years of age
3. Subject is able and willing to give informed consent.

Exclusion Criteria:

1. Patients with known history of atrial arrhythmias.
2. Patients who are not treated with β-blockers unless heart rate is too low for β-blockers assumption.
3. Participation in another clinical trial which may affect the outcome within 3 months prior to day of procedure.
4. Other surgical interventions (e.g. valve replacement) programmed in the same surgical session
5. Resting pulse rate ≤45 beats / min as assessed before daily doses of β-blockage is administered.
6. Hypotension (RR systolic <100 or RR diastolic <50).
7. Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complete bundle branch block.
8. Subject is diagnosed with epilepsy or history of seizures.
9. Coagulation abnormalities as determined by anticoagulation guidelines for neuroaxial procedures 2011.
10. Patients not stabilized on an anti-arrhythmic drug regimen for the last 30 days.
11. Patients with long QT syndrome.
12. Patients with Brugada syndrome.
13. Patients affected by Polyneuropathy (e.g. due to diabetes).
14. Patients affected by pericarditis
15. Patients who underwent procedures in the past, which are expected to have changed the innervation of the heart for example:

    * Ablation procedure
    * Cardiac surgery
16. Pregnant patients or nursing (subjects who are of child bearing potential and are not on a reliable form of birth control will undergo a pregnancy test)
17. Patients already implanted with cardiac devices
18. Patients with existing implanted neurostimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | 5 days after CABG
  AT/AF will be defined as an episode with an atrial rate >175 bpm lasting ≥ 20 seconds.

SECONDARY OUTCOMES:
Medication | 5 days after CABG
  Description of integral medication related to AT/AF occurrence and pain in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery.
Cardioversion | 5 days after CABG
  Description of number of cardioversion needed in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery.
Hospitalizations Days | 1 week after discharge
  Description of hospitalizations longer than 5 days as required by the protocol and clinical practice in the treatment (SCS) and control group.
BP | 5 days after CABG
  Description of 1) intra arterial blood pressure as averaged over the first 24 hours after surgery and 2) arterial blood pressure as determined using a blood pressure cuff at a specific time on Day-2, Day-3, Day-4 and Day-5 after surgery in the treatment (SCS) and control group.
Description of the total number of AT/AF episodes in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery. | 5 days after CABG
  AT/AF episodes
Description of burden of AT/AF episodes in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery. | 5 days after CABG
  AT/AF burden
Premature atrial beats | 5 days after CABG
  Description of the amount of premature atrial beats in the treatment (SCS) and control group from the end of the procedure till Day-5 after surgery.
VT/VF episodes | 5 days after CABG
  Description of the total number of VT/VF episodes in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery.
Burden VT/VF episodes | 5 days after CABG
  Description of the burden of VT/VF episodes in the treatment (SCS) and control group between start of anesthesia and 5 days after surgery.
HRV | 5 days after CABG
  Improvement LF/HF ratio of Heart Rate Variability (HRV) by SCS. SCS On and Off will be compared in each patients in the treatment (SCS) group before surgery and 5 days after surgery.
Pain on the VAS scale | 5 days after CABG
  Description of pain-score due to CABG surgery measured with a VAS score three times a from Day-1 till Day-5 after surgery in the treatment (SCS) and control group.
Bladder function | 5 days after CABG
  The extra time the bladder catheter will be kept in the patients after the first 2 days after surgery will be described in the treatment (SCS) and control group in order to assess bladder function.
HR | 5 days after CABG
  Description of 1) heart rate as averaged over the first 24 hours after surgery and 2) heart rate as determined using a blood pressure cuff at a specific time on Day-2, Day-3, Day-4 and Day-5 after surgery in the treatment (SCS) and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Diephuis, PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente (MST), Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided